CLINICAL TRIAL: NCT05771818
Title: A Community-Based Falls Prevention Program for Adults At-Risk for Falls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UR-0627-320
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Accidental Fall; Neurologic Disorder; Old Age; Debility; Healthy Aging
Keywords: Falls, Balance, Neurological, Geriatrics, Risk
MeSH Terms: conditions — Nervous System Diseases; Frailty; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Falls Prevention training (Experimental): The intervention consists of 10 sessions. One session a week consists of obstacle course training. The other session consists of falls strategies and walking and balance exercises. Each session lasts approximately 1.5 hours
  Interventions: Other: Falls Prevention Program

INTERVENTIONS:
Other: Falls Prevention Program — The intervention consists of 10 sessions. One session a week consists of obstacle course training. The other session focuses on falls strategies training and walking and balance exercises. Each session lasts approximately 1.5 hours.

SUMMARY:
The goal of this interventional study is to implement a Falls Prevention Program to impact the risk and injuries related to falls. The main question is to learn and examine the effects of a falls prevention program on the functional mobility of adults at risk for falls.

Participants will:

* Complete functional mobility assessments
* Complete Falls prevention obstacle course training
* Complete Falls Strategies Training
* Complete walking and balance training

DETAILED DESCRIPTION:
The purpose of the study is to implement a Fall Prevention Program to impact the risk and injuries related to falls. This study is innovative in that (1) it will be implemented as a community service program for the first time in the United States (2) it will attempt to standardize an obstacle course as a reliable and valid outcome measure for balance and falls (3) it will incorporate community outreach learning opportunity for students in a doctor of physical therapy curriculum at the University of St. Augustine for Health Sciences and (4) it will assess effectiveness using a variety of standardized and valid outcome measures to address balance and coordination deficits, fear of falling, incidence of falling, gait speed, feasibility and patient perception and satisfaction.

Specific Aim 1: To examine the effects of a falls prevention program on the functional mobility of adults at risk for falls. Hypothesis: Physical exercise and dynamic balance training has been shown to be effective in decreasing risk for falls. The Falls Prevention Program will have a positive effect on balance, gait speed, fear of falls, incidence of falls and incorporation of falls techniques.

Specific Aim 2: To create a falls prevention program within a Doctor of Physical Therapy curriculum. Hypothesis: Community outreach which are learning opportunities that benefit the community at large are part of the Doctor of Physical Therapy curriculum. It is expected that the Falls Prevention Program will be successfully integrated into the Geriatric Rehabilitation for Physical Therapy course with appropriate participation from the students.

Specific Aim 3: Evaluate the reliability and validity of an obstacle course as a measure of fall risk. Hypothesis: The Falls Prevention Program includes a 17-item obstacle course that significantly challenges the participant's functional mobility and standing dynamic balance. It is expected that the obstacle course will serve as a reliable and valid test for the assessment for balance and mobility.

Specific Aim 4: Evaluate the acceptability of a Falls Prevention Program. Hypothesis: There are no current falls prevention programs available to the community as a free community service program. It is believed that the program will be accepted by the community as well as the faculty and students leading the program.

Specific Aim 5: Determine whether disease moderates the relationship between the effects of a Falls Prevention Program and functional mobility of adults at risk for falls. Hypothesis: Fall Prevention Programs to improve balance and functional mobility have been effective for participants at risk for falls. This program will aim to assess the impact a Falls Prevention Program has on different populations.

Specific Aim 6: Determine the effects of the Falls Prevention Program on Anticipatory Postural Assessment and Compensatory Postural Assessment.

Hypothesis: Older adults will improve their Anticipatory Postural Assessment and Compensatory Postural Assessment (less magnitude and faster responses of muscle activity along with less body displacement) in response to balance perturbations a a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age range: 18-100
* At risk for falls (as determined by any of the following:
* Positive history of falls within 5 years
* Timed up and Go <45 seconds
* Medical clearance for participation in Falls Prevention Program
* Able to attend biweekly sessions for 5 weeks

Exclusion Criteria:

* Unable to independently kneel and sit and on the floor and return to chair
* Taking prescription anti-coagulants without physician clearance to participate
* No medical clearance for participation in Falls Prevention Program
* Unable to attend bi-weekly on-site sessions for 5 weeks
* Other reasons that may limit participation in intervention

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes over time in Activities-Specific Balance Confidence Scale from baseline to one year | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The Activities-Specific Balance Confidence Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness.
Changes in Falls Efficacy Scale - International from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  A self-administered questionnaire designed to assess fear of falling in mainly community-dwelling older population
Changes in Berg Balance Test from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The Berg Balance Test is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks
Changes in Functional Reach Test from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The Functional Reach measures the participant to complete a forward reach while in a standing position
Changes in Single Limb Stance from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The Single Limb Stance test is a measurement to assess the individual's ability to stand unsupported on one limb.
Changes in Tandem Stance from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The Tandem Stance test is a measurement to assess the individual's ability to stand unsupported with one foot directly in front of the other
Changes in 10-Meter Walk Test from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance
Changes in 6-Minute Walk Test from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance
Changes in Timed Up and Go from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The Timed Up and Go test is a measure that assess fall risk by performing sit to stand and walking
Changes in Anticipatory & Compensatory Postural Assessment from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  Electromyography measure of postural stability in standing
Changes in Obstacle Course performance from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The obstacle course measures time to complete 17 obstacles and errors performed on each of the obstacles
Changes in falls occurrences from baseline to 1-year post | Baseline, 6-weeks, 6-months and 1-year post intervention.
  The questionnaire assesses incidence of falls, falls with injuries and falls requiring hospitalization
Changes Physical Activity Intensity Monitoring from baseline to 1-year post intervention | Baseline, 6-weeks, 6-months and 1-year post intervention.
  Heart rate monitoring during all components of falls prevention program

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Garcia, PT, DPT, EdD, Principal Investigator — University of St. Augustine for Health Sciences
Locations (1):
- University of St Augustine for Health Science, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weerdesteyn V, Rijken H, Geurts AC, Smits-Engelsman BC, Mulder T, Duysens J. A five-week exercise program can reduce falls and improve obstacle avoidance in the elderly. Gerontology. 2006;52(3):131-41. doi: 10.1159/000091822. PMID 16645293
- [Result] Rosendahl E, Gustafson Y, Nordin E, Lundin-Olsson L, Nyberg L. A randomized controlled trial of fall prevention by a high-intensity functional exercise program for older people living in residential care facilities. Aging Clin Exp Res. 2008 Feb;20(1):67-75. doi: 10.1007/BF03324750. PMID 18283231
- [Result] Gallo E, Stelmach M, Frigeri F, Ahn DH. Determining Whether a Dosage-Specific and Individualized Home Exercise Program With Consults Reduces Fall Risk and Falls in Community-Dwelling Older Adults With Difficulty Walking: A Randomized Control Trial. J Geriatr Phys Ther. 2018 Jul/Sep;41(3):161-172. doi: 10.1519/JPT.0000000000000114. PMID 27893567
- [Result] Hewitt J, Goodall S, Clemson L, Henwood T, Refshauge K. Progressive Resistance and Balance Training for Falls Prevention in Long-Term Residential Aged Care: A Cluster Randomized Trial of the Sunbeam Program. J Am Med Dir Assoc. 2018 Apr;19(4):361-369. doi: 10.1016/j.jamda.2017.12.014. PMID 29402651
- [Result] Gudnadottir M, Thorsteinsdottir TK, Mogensen B, Aspelund T, Thordardottir EB. Accidental injuries among older adults: An incidence study. Int Emerg Nurs. 2018 Sep;40:12-17. doi: 10.1016/j.ienj.2018.03.003. Epub 2018 Apr 13. PMID 29661594
- [Result] Stewart Williams J, Kowal P, Hestekin H, O'Driscoll T, Peltzer K, Yawson A, Biritwum R, Maximova T, Salinas Rodriguez A, Manrique Espinoza B, Wu F, Arokiasamy P, Chatterji S; SAGE collaborators. Prevalence, risk factors and disability associated with fall-related injury in older adults in low- and middle-incomecountries: results from the WHO Study on global AGEing and adult health (SAGE). BMC Med. 2015 Jun 23;13:147. doi: 10.1186/s12916-015-0390-8. PMID 26099794
- [Result] Oyetunji TA, Ong'uti SK, Bolorunduro OB, Gonzalez DO, Cornwell EE, Haider AH. Epidemiologic trend in elderly domestic injury. J Surg Res. 2012 Apr;173(2):206-11. doi: 10.1016/j.jss.2011.05.003. Epub 2011 May 31. PMID 21704329
- [Result] Saveman BI, Bjornstig U. Unintentional injuries among older adults in northern Sweden--a one-year population-based study. Scand J Caring Sci. 2011 Mar;25(1):185-93. doi: 10.1111/j.1471-6712.2010.00810.x. PMID 20626698
- [Result] Scariot V, Rios JL, Claudino R, Dos Santos EC, Angulski HBB, Dos Santos MJ. Both anticipatory and compensatory postural adjustments are adapted while catching a ball in unstable standing posture. J Bodyw Mov Ther. 2016 Jan;20(1):90-97. doi: 10.1016/j.jbmt.2015.06.007. Epub 2015 Jun 19. PMID 26891642